CLINICAL TRIAL: NCT00651287
Title: A 12-Week Open-Label, Uncontrolled Multicenter Study to Assess the Efficacy and Safety of Quinapril or Quinapril Plus Hydrochlorothiazide in Subjects With Mild to Moderate Hypertension
Brief Title: A Study to Evaluate the Efficacy and Safety of Quinapril or Quinapril Plus Hydrochlorothiazide in Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A9061007
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Quinapril; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- quinapril 20 mg (Active Comparator)
  Interventions: Drug: quinapril 20 mg
- quinapril 20 mg+hydrochlorothiazide 12.5 mg (Active Comparator)
  Interventions: Drug: quinapril 20 mg plus hydrochlorothiazide 12.5 mg
- quinapril 40 mg (Active Comparator)
  Interventions: Drug: quinapril 40 mg

INTERVENTIONS:
Drug: quinapril 20 mg — Quinapril 20 mg oral tablet daily for the first 6 weeks, and if a responder, continued on quinapril 20 mg for an additional 6 weeks
  Arms: quinapril 20 mg
Drug: quinapril 20 mg plus hydrochlorothiazide 12.5 mg — Quinapril 20 mg oral tablet daily for the first 6 weeks; if nonresponder, could be randomized to quinapril 20 mg plus hydrochlorothiazde 12.5 mg daily (Accuzide tablets) for 6 weeks
  Arms: quinapril 20 mg+hydrochlorothiazide 12.5 mg
Drug: quinapril 40 mg — Quinapril 20 mg oral tablet daily for the first 6 weeks; if nonresponder, could be randomized to quinapril 40 mg oral tablet daily for 6 weeks
  Arms: quinapril 40 mg

SUMMARY:
The purpose of this study is to determine the response rate for the therapeutic goal (diastolic blood pressure (BP) less than 90 mmHg and systolic BP less than 140 mmHg) at Week 6 for quinapril 20 mg and at Week 12 for quinapril 20 mg, quinapril 40 mg, and quinapril 20 mg plus hydrochlorothiazide 12.5 mg; and to determine the mean decrease in diastolic and systolic BP measurements and the change in heart rate at Week 6 and Week 12 compared with baseline.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of mild to moderate primary hypertension ("Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure, 6th report" Stage I or II)
* Sitting diastolic blood pressure between 90 mmHg and 109 mmHg and systolic blood pressure between 140 mmHg and 179 mmHg at the end of the no-treatment run-in period

Exclusion Criteria:

* Subjects with secondary hypertension
* Subjects with serious cardiac disease (including myocardial infarction in the last 3 months or decompensated heart failure)
* Subjects who do not accept to stop using any other antihypertensive treatment during the run-in period and the treatment period of the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2002-12; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Response rate for the therapeutic goal (at Week 6 for 20mg quinapril and at Week 12 for 40mg quinapril and 20mg quinapril plus 12.5mg hydrochlorothiazide) | 12 weeks

SECONDARY OUTCOMES:
Mean decrease in diastolic and systolic BP measurements at Week 6 and at Week 12 compared to baseline | 12 weeks
Change in heart rate at Week 6 and at Week 12 compared to baseline | 12 weeks
Adverse events were recorded throughout the study | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Cerrahpaşa, Istanbul
  - Pfizer Investigational Site, Diyarbak R
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9061007&StudyName=A%20Study%20to%20Evaluate%20the%20Efficacy%20and%20Safety%20of%20Quinapril%20or%20Quinapril%20Plus%20Hydrochlorothiazide%20in%20Patients%20with%20Mild%20to%20Moderate%20Hyper